CLINICAL TRIAL: NCT03837262
Title: GLucose Monitoring Programme SingaporeE (GLiMPSE) - Phase 1
Brief Title: GLucose Monitoring Programme SingaporeE (GLiMPSE)
Acronym: GLiMPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: KK Women's and Children's Hospital (Other Government); SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GLiMPSE-POC1
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Flash Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Feasibility study assessing the use of flash glucose monitoring together with structured education to improve outcomes in Type 2 diabetes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Flash glucose monitoring (Experimental): Flash glucose monitoring continuously for 6 weeks then once a month up to 24 weeks, with structured education
  Interventions: Combination Product: Flash Glucose Monitoring and structured education

INTERVENTIONS:
Combination Product: Flash Glucose Monitoring and structured education — A feasibility study assessing the use of flash glucose sensing technology with structured education to improve glycemic outcomes in T2D adults and children

SUMMARY:
This phase 1 study is a non-randomized, single-arm, multi-center study that is designed to evaluate the feasibility and acceptability of the flash glucose monitoring system together with a structured education programme in individuals with Type 2 Diabetes.

DETAILED DESCRIPTION:
Up to 30 adults and 15 children will be recruited from 3 different sites in Singapore.

For Adults, this phase consists of screening and intervention periods.

Screening Period (Week -2 to -1):

Participants will be asked to wear a blinded flash glucose monitoring system and will be asked to continue testing their capillary glucose readings at least once daily for 2 weeks (week -2 to week -1). Sensor glucose measurements are not available to both participants and investigators during this screening period. Participants who are able to wear the sensor for the 2 weeks, and are monitoring their capillary glucose levels at least 70% of the time for the 2 weeks (>10 readings/2weeks), will proceed on with the intervention period.

Intervention Period (Week 0 - 26):

Participants will wear a personal version of the flash glucose monitoring system continuously for the next 6 weeks. After these 6 weeks, they will wear the sensor intermittently (one sensor lasting 2 weeks, per 4 weeks) for the following 18 weeks.Participants in this arm will receive an education package that consists of Diabetes nurse educator and/or dietitian appointments during weeks 0, 2, 6 and 24. After week 24, they will put on a blinded sensor for the last 2 weeks of the intervention period (week 25 to week 26). HbA1c will be monitored at weeks 0, 14 and 24. Questionnaires will be administered to assess acceptability of wear, and perceived value to the end-user.

Paediatric participants will not undergo blinded sensor wear but will undergo the intervention period, with the schedule of wear identical to the adults'. The education curriculum will be age-appropriate and will be delivered over weeks 0, 2, 6, 12, and 24. Their HbA1c will be monitored at week 0, 12 and 24. Questionnaires will be administered to assess acceptability of wear, and perceived value to the end-user.

ELIGIBILITY:
Inclusion Criteria:

Adults

1. Adults (Age > 21 years) with Type 2 diabetes (HbA1c 8 to 10% at time of enrolment)
2. Singapore Citizen or Permanent Resident
3. Treatment with diet and exercise alone or other glucose-lowering therapies except prandial insulin. GLP-1 agonists and / or basal insulin (NPH insulin, Insulin Lantus, Insulin Toujeo, Insulin Detemir) are permitted.
4. Self-reported regular blood glucose testing via CBG (more than 3/week)

Children

1. Children and adolescents (Age between 12 and 21 years old) with Type 2 diabetes and HbA1c >8% at the time of enrolment
2. Singapore Citizen or Permanent Resident
3. Insulin replacement as part of diabetes management

Exclusion Criteria:

1. Age above 75 years
2. Type 1 diabetes, monogenic diabetes
3. Prandial insulin (quick-acting insulin or premixed insulin)
4. Cancer requiring treatment in the past 5 years
5. Chronic renal failure (eGFR<45ml/min) or dialysis
6. Amputation of lower limbs (excluding toe amputations)
7. Bariatric surgery for weight loss
8. Current systemic treatment with steroids
9. Pregnancy, attempting pregnancy or lactation.
10. Haemolytic anaemia or haemoglobinopathy
11. Prior use of the flash glucose monitoring system

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention | 26 weeks
  Record of the number of subjects screened, enrolled and subsequently retained through the 26 weeks of follow up at 3 sites

SECONDARY OUTCOMES:
Questionnaire | 24 weeks
  Questionnaire to assess the acceptability of wear of the flash glucose monitoring system
HbA1c | 24 weeks
  Measurement of HbA1c will be performed at baseline, week 12 and week 24
DSS questionnaire | 24 weeks
  Diabetes Distress scale to be administered at baseline and week 24
EQ-5D-5L Questionnaire | 24 weeks
  EQ-5D-5L Questionnaire to be administered at baseline and week 24
WPAI questionnaire | 24 weeks
  Work Productivity and Activity impairment questionnaire to be administered at baseline and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Daphne SL Gardner, MD, Principal Investigator — Singapore General Hospital, SingHealth
Locations (3):
- Singapore (3):
  - Singapore General Hospital, Singapore
  - KKH, Singapore
  - Pasir Ris Polyclinic, Singapore

IPD SHARING:
Plan to Share IPD: Undecided